CLINICAL TRIAL: NCT03718676
Title: Clinical and Radiographic Comparison of RetroMTA, OrthoMTA And Ferric Sulfate for Pulpotomy in Primary Molars
Brief Title: Pulpotomy With Various MTA Materials and Ferric Sulphate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Sultan KELES, Assist. Prof.Dr., Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-047
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2018-10

CONDITIONS: Pulpotomy
Keywords: pulpotomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ferric sulphate (Other): Group FS. Teeth in this goup will pulpotomized with ferris-sulphate.
  Interventions: Procedure: Ferric sulphate
- Orto-mta (Experimental): Group O-MTA.Teeth in this goup will pulpotomized with Ortho-mta.
  Interventions: Procedure: Ortho-MTA
- Retro-mta (Experimental): Group R-MTA. Teeth in this goup will pulpotomized with Retro-mta.
  Interventions: Procedure: Retro-MTA

INTERVENTIONS:
Procedure: Ferric sulphate — Teeth were pulpotomized with ferric sulphate in this group.
  Arms: Ferric sulphate
Procedure: Ortho-MTA — Teeth were pulpotomized with Ortho-MTA in this group.
  Arms: Orto-mta
Procedure: Retro-MTA — Teeth were pulpotomized with Retro-MTA in this group.
  Arms: Retro-mta

SUMMARY:
The aim of this study was to determine clinical and radiographic efficacy of the newly developed OrthoMTA and RetroMTA , compared frequently used ferric sulfate for pulpotomy in primary second molars.

DETAILED DESCRIPTION:
A total of 96 second primary second molars from 32 children ,who met inclusion criteria and were 5-9 years old were selected for the study. Teeth were randomly divided into three groups according to the planned treatment: O-MTA (n=32 teeth), R-MTA (n=32 teeth) and FS (n=32 teeth). Clinical and radiographical follow-up examinations were conducted at 3, 6 and 9 months postoperatively. The data were evaluated with Chi-square test, Cochran Q test, Post-Huc Dunn test and Kaplan-Meier analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients have at least three deep carious primary second molars
* Teeth with no spontaneous pain
* Patient who are willing to participate
* Cooperative children

Exclusion Criteria:

* Patients who are not willing to participate
* History of systemic disease
* Pathological mobility
* Presence of internal or external root resorption
* Presence of apical radiolucency

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Clinical success rate | Change of clinical success from Baseline at 18 months
  Clinical success

CONTACTS AND LOCATIONS:
Overall Officials: sultan keles, Dr., Principal Investigator — Pediatric dentistry
Locations (1):
- Sultan KELES, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We will share the results.

REFERENCES:
- [Background] Awawdeh L, Al-Qudah A, Hamouri H, Chakra RJ. Outcomes of Vital Pulp Therapy Using Mineral Trioxide Aggregate or Biodentine: A Prospective Randomized Clinical Trial. J Endod. 2018 Nov;44(11):1603-1609. doi: 10.1016/j.joen.2018.08.004. Epub 2018 Oct 3. PMID 30292451